CLINICAL TRIAL: NCT03761004
Title: A Phase 1 Single-Dose, Open-label, Sequential, Three-Period Crossover Study to Evaluate the Pharmacokinetics of WD-1603 Tablets in Healthy Subjects
Brief Title: WD-1603 PK Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hong Kong WD Pharmaceutical Co., Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WD-1603-1001
Record Dates: First submitted 2018-11-26; First posted 2018-12-03 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- WD-1603 single dose (Experimental): WD-1603 single dose:
  A single WD-1603 tablet after breakfast. Plasma samples for PK analysis will be collected at pre-dose (baseline) and 10 min, 30 min, 45 min and 1, 1.5, 2, 3, 4, 5, 5.5, 6, 7, 8, 10, 12, 16 and 24 hours post-dose.
  Interventions: Drug: carbidopa-levodopa
- WD-1603 BID dose (Experimental): WD-1603 BID dose:
  A single WD-1603 tablet after breakfast, and a second WD-1603 tablet approximately 3 hours after completing lunch.
  Plasma samples for PK analysis will be collected at pre-dose (baseline) and 10 min, 30 min, 45 min and 1, 1.5, 2, 3, 4, 4.5, 5, 6, 7, 7.25, 7.5, 7.75, 8, 8.5, 9, 10, 10.5 11, 12, 16 and 24 hours post-dose.
  Interventions: Drug: carbidopa-levodopa
- Sinemet single dose (Active Comparator): Sinemet single dose:
  A single oral dose of Sinemet after breakfast. Plasma samples for PK analysis will be collected at pre-dose (baseline) and 10 min, 30 min, 45 min and 1, 1.5, 2, 3, 4, 6, 7, 8, 10, 12, 16 and 24 hours post-dose.
  Interventions: Drug: carbidopa-levodopa

INTERVENTIONS:
Drug: carbidopa-levodopa — single dose of WD-1603, BID dose of WD-1603 and Sinemet IR

SUMMARY:
This is a pilot study to investigate if the extended release formulation of WD-1603 generates anticipated plasma concentration profile. The study is an open-label, sequential, 3-way crossover study to evaluate if WD-1603 generates anticipated plasma levodopa exposure compared to Sinemet IR tablets in healthy subjects. The study comprises of a medical Screening visit, three 2-night (3-day) Treatment periods, 2 outpatient visits, and a Follow-up visit. Study drug administration in each Treatment period is separated by a washout interval of 5 days. The Follow-up visit will occur approximately 7 days (±1) following the last study drug administration. The duration of subject participation, including screening, is approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female subjects, 18 to 55 years of age, inclusive, at the time of signing the informed consent form (ICF).
2. A minimum body weight of 50.0 kg (110.0 lbs) and body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive, at screening.
3. Non-smoker for at least 3 months and tests negative on urine cotinine test.
4. Medically healthy subjects with clinically insignificant screening and Day -1 admission results (medical history, 12-lead electrocardiogram (ECG), physical examination, vital signs, and laboratory tests) as determined by the Investigator or designee.
5. Female subjects of childbearing potential with male sexual partners must be using and willing to continue using medically acceptable contraception (true abstinence, hormonal contraceptives [combined oral pill, patch, or vaginal ring], intrauterine device, or double-barrier methods [condom with spermicide, diaphragm or cervical cap with spermicide]) from Screening (or at least 3 months prior to Screening for hormonal contraceptives) until at least 28 days after the last study drug administration.
6. Female subjects of non-childbearing potential must be either post-menopausal (post-menopausal is defined as being amenorrheic for at least 1 year without another cause and a follicle-stimulating hormone [FSH] level ≥26 IU/L) or surgically sterile (hysterectomy, bilateral oophorectomy, or bilateral tubal ligation).
7. Male subjects with female sexual partners of childbearing potential must be using and willing to continue using medically acceptable contraception (true abstinence, vasectomy, or male condom for subjects plus an additional method of contraception for their female partners) from Screening until 28 days following the last administration of study drug.
8. Subjects are able to understand English and to give their signed informed consent before any study-related procedures are performed.

Exclusion Criteria:

1. History of serious allergic reaction or hypersensitivity to levodopa or carbidopa.
2. Subjects with, or a history of, narrow-angle glaucoma, cancer, diabetes, or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, hematologic, dermatological, neurological, psychiatric, or other major disorder.
3. History of clinically significant drug and/or food allergies as determined by the Investigator or designee, or previous status asthmaticus.
4. Subject is not willing to abstain from alcohol for 48 hours prior to admission in Day-1 until the final blood draw is complete through the final day of blood draws.
5. Use of prescription or non-prescription drugs, including herbal and dietary supplements, within 7 days prior to the first dose of study medication.
6. Treatment with an investigational drug within 30 days prior to the first dosing, or more than 5 half-lives of the compound which the subject was treated with , whichever is longer.
7. Donation or loss of more than 500 mL whole blood within 30 days preceding the first dose. Subjects must not donate blood or plasma during the study and for at least 56 days after the Follow-up visit.
8. Difficulty with venous access or unsuitable or unwilling to undergo catheter insertion.
9. Self-reported substance or alcohol dependence (excluding nicotine and caffeine) within the past 2 years prior to dosing, and/or has ever participated or plans to participate in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence.
10. Typical weekly alcohol consumption of 14 alcoholic drinks. One standard alcoholic drink is equivalent to 43 mL (1.5 oz.) hard liquor or 142 mL (5 oz.) wine or 341 mL (12 oz.) beer.
11. Positive results in any of the serology tests of human immunodeficiency virus (HIV) and hepatitis B and C infections.
12. Female subjects who are currently pregnant (have a positive pregnancy test) or lactating or who are planning to become pregnant within 30 days of the last study drug administration.
13. Positive urine drug at Screening and Day -1 admission. Given the long half-life of tetrahydrocannabinol (THC) and its metabolites, subjects with a positive result for THC at Screening may be included at the discretion of the investigator.
14. Positive breath alcohol test. Subjects with a positive result at Screening may be rescheduled at the investigator's discretion.
15. Any condition that, in the opinion of the Investigator or designee, would complicate or compromise the study or the well-being of the subject.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Cmax | pre-dose（baseline）and specified time points up to 24 hours post-dose(as specified in the Arm/Group description)
  the maximum plasma concentrations
AUC0-t | pre-dose（baseline）and specified time points up to 24 hours post-dose(as specified in the Arm/Group description)
  the areas under the plasma concentration versus time curve calculated from 0 to the last measurable observation
AUC0-inf | pre-dose（baseline）and specified time points up to 24 hours post-dose(as specified in the Arm/Group description)
  the areas under the plasma concentration versus time curve extrapolated from 0 to infinity

CONTACTS AND LOCATIONS:
Locations (1):
- INC Research Toronto, Inc., Toronto, Canada